CLINICAL TRIAL: NCT05654532
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Anti-Tumor Activity of AC699 in Patients With Estrogen Receptor Positive/Human Epidermal Growth Factor Receptor 2 Negative (ER+/HER2-) Locally Advanced or Metastatic Breast Cancer
Brief Title: Study of AC699 in Patients With Estrogen Receptor Positive/Human Epidermal Growth Factor Receptor 2 Negative (ER+/HER2-) Locally Advanced or Metastatic Breast Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Accutar Biotechnology Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AC699-001
Record Dates: First submitted 2022-12-08; First posted 2022-12-16 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Estrogen receptor-positive breast cancer; ER positive; ER+; Human epidermal growth factor receptor 2 negative; HER2 negative breast cancer; HER2-; AC699; Metastatic breast cancer; MBC; Locally advanced breast cancer; ER chimeric degrader; ER degrader
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AC699 Dose Escalation (Experimental): Participants will receive an assigned dose of AC699 monotherapy during dose escalation.
  One cycle is defined as 28 days.
  Interventions: Drug: AC699

INTERVENTIONS:
Drug: AC699 — Participants will receive AC699 orally daily in 28-day cycles.

SUMMARY:
This clinical trial is evaluating a drug called AC699 in participants with estrogen receptor positive/human epidermal growth factor 2 negative (ER+/HER2-) locally advanced or metastatic breast cancer. The main goals of this study are to:

* Identify the recommended dose of AC699 that can be given safely to participants
* Evaluate the safety profile of AC699
* Evaluate the pharmacokinetics of AC699
* Evaluate the effectiveness of AC699

DETAILED DESCRIPTION:
This study is a Phase I, first-in-human, open-label dose-escalation study of AC699, an orally bioavailable estrogen receptor degrader, given as a single agent.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent (ICF)
* Adult male and female participants, at least 18 years-of-age at the time of signature of the ICF
* Female participants must be postmenopausal
* Confirmed diagnosis of advanced, unresectable, and/or metastatic breast cancer following disease progression on standard treatment, or for whom no therapy of proven efficacy exists, or who are not amenable to standard therapies
* Histologically and/or cytologically confirmed diagnosis of estrogen-receptor positive (ER+) human epidermal growth factor 2 negative (HER2-) breast cancer
* Must have received at least 2 prior endocrine or at least 1 prior line of endocrine therapy if combined with CDK4/6 inhibitor
* Prior chemotherapy is not required, but up to 3 prior regimens of cytotoxic chemotherapy will be allowed in the locally advanced/ metastatic setting
* At least 1 measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 (Appendix B) or at least 1 predominantly lytic bone lesion in the absence of measurable disease
* Acceptable organ and hematologic function at baseline
* Life expectancy ≥12 weeks after the start of the treatment

Exclusion Criteria:

* Treatment with any of the following:

  * Any cytotoxic chemotherapy, investigational agents or other anti-cancer drugs for the treatment of locally advanced or metastatic breast cancer within 14 days prior to the first administration of AC699
  * Radiation therapy within 14 days prior to first study drug administration that did not resolve to tolerable toxicity, or prior irradiation to >25% of bone marrow. Prior palliative radiotherapy to metastatic lesion(s) is permitted, provided it has been completed 7 days prior to study enrollment and no clinically significant toxicities are expected (e.g., mucositis, esophagitis).
  * Major surgery within 21 days prior to the first study drug administration (exception: participants may enroll if fully recovered or without intolerable or clinically significant adverse effects but at least 14 days must have elapsed between major surgery and first study drug administration)
* Known symptomatic brain metastases requiring the use of systemic corticosteroids ≥10 mg/day prednisone or equivalents. Asymptomatic and treated, or asymptomatic untreated brain metastases are allowed as long as participants are clinically stable. Stable doses of anticonvulsants are allowed.
* Any condition that impairs a participant's ability to swallow whole pills. Impairment of gastrointestinal function (GI) or GI disease or other condition at baseline that will interfere significantly with the absorption, distribution, or metabolism of AC699.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-12-29 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (DLTs) from AC699 monotherapy | First 28 days of treatment. Cycles are 28 days.
Incidence of treatment-emergent adverse events (TEAEs) and clinically significant Grade 3 or higher lab abnormalities following administration of AC699 | Approximately 18 months.

SECONDARY OUTCOMES:
Objective response rate (ORR) to assess the anti-tumor activity of AC699 | Approximately 18 months.
Clinical Benefit Rate (CBR) to assess the anti-tumor activity of AC699 using RECIST 1.1 | Approximately 18 months.
Duration of Response (DOR) to assess the anti-tumor activity of AC699 using RECIST 1.1 | Approximately 18 months.
Disease Control Rate (DCR) to assess the anti-tumor activity of AC699 using RECIST 1.1 | Approximately 18 months.
Progression Free Survival (PFS) to assess the anti-tumor activity of AC699 using RECIST 1.1 | Approximately 18 months.
Pharmacokinetic Analysis: Area under the concentration-time curve over the dosing interval (AUC(0-infinity)) | Up to approximately 28 weeks
Pharmacokinetic Analysis: Area under the concentration-time curve over the dosing interval (AUC(0-tau)) | Up to approximately 28 weeks
Pharmacokinetic Analysis: Maximum plasma concentration (Cmax) | Up to approximately 28 weeks
Pharmacokinetic Analysis: Time to maximum plasma concentration (tmax) | Up to approximately 28 weeks
Pharmacokinetic Analysis: Terminal elimination half-life (t1/2) | Up to approximately 28 weeks

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Site 08, Denver, Colorado
  - Site 07, Orlando, Florida
  - Site 02, Sarasota, Florida
  - Site 06, Rockville, Maryland
  - Site 01, Nashville, Tennessee
  - Site 03, Houston, Texas
  - Site 09, San Antonio, Texas
  - Site 05, Norfolk, Virginia
  - Site 04, Vancouver, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hamilton E, Layman RM, Cosgrove D, Danso M, Zhang H, He W, Kim SY, Fan J, Patel MR. ER degradation for ER+/HER2- advanced or metastatic breast cancer: a phase 1 trial. Nat Commun. 2025 Dec 17. doi: 10.1038/s41467-025-67485-y. Online ahead of print. PMID 41407710